CLINICAL TRIAL: NCT01390597
Title: The Molecular Mechanisms of Transformation in Peripheral T-cell and NK Lymphomas
Brief Title: Biomarkers in Tumor Tissue Samples From Patients With Peripheral T-cell Lymphoma or Natural Killer Cell Neoplasms
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000703260; ECOG-E2404T1
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: peripheral T-cell lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Peripheral; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Cytogenetic Analysis; Chromosome Mapping; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA analysis
Genetic: cytogenetic analysis
Genetic: gene mapping
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat the cancer.

PURPOSE: This research trial studies biomarkers in tumor tissue samples from patients with peripheral T-cell lymphoma or natural killer cell neoplasms.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify mutations in oncogenes and tumor suppressors of peripheral T-cell lymphoma or natural killer (NK) cell neoplasm.
* To delineate the mechanisms that mediate oncogenic effects and their clinical prognostic significance in these diseases.
* To perform a comprehensive mutation analysis via whole exome resequencing in a panel of peripheral T-cell or NK lymphomas.

OUTLINE: Fixed paraffin-embedded tumor tissue samples are analyzed for mutations by the Illumina HiSeq platform. Sequencing reads are performed by GAPipeline version 1.5.1 and mapping on the human genome performed using the MAQ software version 0.7.1. Genes harboring validated somatic mutations are then amplified by PCR and analyzed by Sanger resequencing.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with peripheral T-cell lymphoma or natural killer cell neoplasms
* Available fresh tumor samples from patients treated on ECOG-E2404 and normal DNA (non-ECOG) samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patient enrolled on E2404 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2011-08-28 (Actual); Study Completion 2011-08-28 (Actual)

PRIMARY OUTCOMES:
New somatically mutated genes in T-cell and NK lymphoma samples | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo A. Ferrando, MD, PhD, Principal Investigator — Herbert Irving Comprehensive Cancer Center